CLINICAL TRIAL: NCT04761627
Title: A Multicenter, Randomized, Double-blinded Study Evaluating the Pharmacokinetics, Efficacy and Safety of Multiple Switches Between Ustekinumab and ABP 654 Compared With Continued Use of Ustekinumab in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Investigate Interchangeability of ABP 654 for the Treatment of Participants With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20200417; 2020-005205-42 (EudraCT Number)
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Psoriasis
Keywords: Psoriasis; Biosimilar; Psoriasis area and severity index; Ustekinumab; Skin Diseases; Dermatologic Agents; Papulosquamous
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The investigators, study personnel (with the exception of the Data Monitoring Committee (DMC), and unblinded Parexel staff supporting DMC activities and randomization list activities) and the study participants will remain blinded to treatment allocation. ABP 654 and ustekinumab will be coded and labeled in a manner that protects blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continued-use Group (Ustekinumab) (Active Comparator): Participants will receive subcutaneous injection of ustekinumab up to Week 52.
  Interventions: Drug: Ustekinumab
- Switching Group (Ustekinumab - ABP 654) (Experimental): Participants will initially receive injection of ustekinumab up to Week 16. Thereafter, starting from Week 28, participants will switch between ABP 654 and ustekinumab every 12 weeks up to Week 52.
  Interventions: Drug: Ustekinumab; Drug: ABP 654

INTERVENTIONS:
Drug: Ustekinumab — Participants will receive subcutaneous (SC) injection of ustekinumab.
  Other Names: Stelara®
Drug: ABP 654 — Participants will receive SC injection of ABP 654.
  Arms: Switching Group (Ustekinumab - ABP 654)

SUMMARY:
The purpose of the study is to evaluate pharmacokinetic similarity, efficacy, safety and immunogenicity of multiple switches between ustekinumab and ABP 654 compared with continued use of ustekinumab in participants with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a multi-center study and will enroll approximately 480 participants.

After eligibility confirmation, all participants will be randomized in a 1:1 ratio into 2 treatment arms: continued use of ustekinumab or multiple switches between ustekinumab and ABP 654 at Week 28. The randomization will be stratified by prior biologic use for psoriasis (yes versus [vs] no) at baseline (Week 0), geographic region, and baseline (Week 0) body weight.

All participants will receive an initial 3 doses of ustekinumab on Day 1 (Week 0), Week 4 and Week 16. At Week 28, participants will be randomized to continue on ustekinumab or switching between ABP 654 and ustekinumab every 12 weeks.

At Week 28, efficacy assessments will be conducted including evaluation of Psoriasis and Area Severity Index (PASI). Participants who do not achieve PASI 50 response or better improvement at Week 28 will be considered as run-in failures and will not be randomized at Week 28; these participants will complete End of Study procedures at Week 28. The run-in period will occur from Day 1 until randomization at Week 28. Those unable to complete the Week 28 visit or did not have a PASI assessment completed at Week 28 will be discontinued from the study.

The total duration of study participation for each participant will be 68 weeks, with up to 4 weeks for screening and 64 weeks after the first investigational product administration.

ELIGIBILITY:
Inclusion Criteria:

* Participant has stable moderate to severe plaque psoriasis for at least 6 months
* Participant has a score of PASI ≥ 12, involvement of ≥ 10% body surface area and static Physician Global Assessment ≥ 3 at screening and at baseline
* Participant is a candidate for phototherapy or systemic therapy
* Participant has previous failure, inadequate response, intolerance, or contraindication to at least 1 conventional antipsoriatic systemic therapy
* Female participant should have a negative serum pregnancy test during screening and a negative urine pregnancy test at baseline
* Participant or legally acceptable representative is capable of giving signed Institutional Review Board (IRB)/Independent Ethics Committee (IEC) informed consent
* Participant has no known history of latent or active tuberculosis
* Participant with a positive purified protein derivative (PPD) test and a history of Bacillus Calmette-Guérin (BCG) vaccination is allowed with a negative Quantiferon/T-spot test
* Participant with a positive PPD test or participant with a positive or indeterminate Quantiferon/T-spot test is allowed if he/she has all the following:

  * No symptoms per tuberculosis worksheet provided by the sponsor, Amgen Inc.
  * Documented history of adequate prophylaxis initiation prior to receiving investigational product in accordance with local recommendations
  * No known exposure to a case of active tuberculosis after most recent prophylaxis
  * No evidence of active tuberculosis on chest radiograph within 3 months prior to the first dose of investigational product

Exclusion Criteria:

* Participant has erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication induced psoriasis, or other skin conditions at the time of screening (eg, eczema) that would interfere with evaluations of the effect of investigational product of psoriasis
* Participant has an active infection or history of infections
* Participant has uncontrolled, clinically significant systemic disease, such as uncontrolled diabetes mellitus, cardiovascular disease, renal disease, liver disease, or hypertension
* Participant has a mean QT internal or abnormal long QT syndrome corrected using Fridericia's formula (QTcF) of > 450 msec (for male participant) or > 470 msec (for female participant) at baseline that, in the opinion of the Investigator, is abnormal or clinically significant
* Participant has moderate to severe heart failure (New York Heart Associate class III/IV)
* Participant has known hypersensitivity to the investigational product or to any of the excipients
* Participant has laboratory abnormalities at screening
* Participant has had previous treatment with any agent specifically targeting interleukin (IL)-12 or IL-23 within 1 year prior to enrollment
* Participant has received biologic treatment for psoriasis within the previous month or 5 drug half-lives (whichever is longer) prior to enrollment
* Participant has received any investigational agents within the previous month or 5 half-lives (whichever is longer) prior to enrollment
* Participant has received non-biologic systemic psoriasis therapy within 4 weeks prior to enrollment
* Participant has received ultraviolet A phototherapy (with or without psoralen) or excimer laser within 4 weeks prior to enrollment, or ultraviolet B phototherapy within 2 weeks prior to enrollment
* Participant has received topical psoriasis treatment within 2 weeks prior to enrollment
* Participant has received other investigational procedures within 4 weeks prior to enrollment and during the course of the study
* Female participant is pregnant or breastfeeding or planning to become pregnant while participating in the study and for at least 5 months after the last dose of investigational product
* Sexually active participants and their partners who are of childbearing potential and not agreeing to use adequate protocol defined contraception methods while participating in the study and for 5 months after the last dose of investigational product

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (88):
- United States (31):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Zenith Research Inc., Beverly Hills, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Quest Dermatology Research, Northridge, California
  - Southern California Dermatology, Inc, Santa Ana, California
  - Encore Research Group-Jacksonville Center for Clinical Resea, Jacksonville, Florida
  - Altus Research, Inc., Lake Worth, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Leavitt Medical Associates of Florida d/b/a Ameriderm Research, Ormond Beach, Florida
  - Riverchase Dermatology and Cosmetic Surgery, Pembroke Pines, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Hamilton Research, LLC, Alpharetta, Georgia
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Dundee Dermatology, West Dundee, Illinois
  - DS Research, Clarksville, Indiana
  - Integrated Clinical Trial Services Inc., West Des Moines, Iowa
  - Kansas Medical Clinic, PA, Topeka, Kansas
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Skin Specialists PC, Omaha, Nebraska
  - ActivMed Practices & Research, LLC., Portsmouth, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - The Dermatology Group, PC, Verona, New Jersey
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Oregon Medical Research Center, Portland, Oregon
  - Austin Institute for Clinical Research, Inc., Dripping Springs, Texas
  - Austin Institute for Clinical Research, Inc - Dermatology, Pflugerville, Texas
  - Progressive Clinical Research [Texas], San Antonio, Texas
  - Center for Clinical Studies, LTD., LLP, Webster, Texas
- Canada (14):
  - Enverus Medical Research, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Dr. Irina Turchin PC Inc., Fredericton, New Brunswick
  - CCA Medical Research, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - Dr Wei Jing Loo Medicine Professional Corporation, London, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - DermEdge Research Inc., Mississauga, Ontario
  - Dr. S. K. Siddha Medicine Professional Corporation - Doctor's Office, Newmarket, Ontario
  - North York Research Inc. - Dermatology, North York, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario
  - Research Toronto, Toronto, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
- Estonia (4):
  - Confido Private Medical Clinic - General Practice/Medicine, Tallinn, Harju
  - Clinical Research Center, Tartu, Tartu
  - Tartu University Hospital, Tartu, Tartu
  - Innomedica OÜ, Tallinn
- Georgia (5):
  - Acad.Fridon Todua Medical Center- Research Institute of Clinical Medicine, Tbilisi, K'alak'i T'bilisi
  - LTD Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi, K'alak'i T'bilisi
  - ,,Tbilisi Cancer center"LTD, Tbilisi, K'alak'i T'bilisi
  - LTD Aversi Clinic, Tbilisi, K'alak'i T'bilisi
  - ,,KANVENI - Scientific/Research National Center of Dermatology and Venereology LLC, Tbilisi
- Germany (11):
  - Derma-Study-Center-FN, Friedrichshafen, Baden-Wurttemberg
  - Dermazentrum Augsburg, Augsburg, Bavaria
  - Dermatologische Gemeinschaftspraxis Dres.Scholz Sebastian Schilling, Mahlow, Brandenburg
  - Universitätsklinikum Frankfurt am Main - Klinik für Dermatol, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Praxis Hoffmann, Witten, North Rhine-Westphalia
  - Klinische Forschung Dresden GmbH, Dresden, Saxony
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - UK-SH - Lübeck, Lübeck, Schleswig-Holstein
  - Charite - Campus Charite Mitte (CCM) - Dermatologie & Allergologie - Dermatologie & Allergologie, Berlin
  - Rothhaar Studien GmbH, Berlin
- Hungary (4):
  - Debreceni Egyetem Klinikai Központ Nagyerdei Campus, Debrecen, Hajdú-Bihar
  - Brgyógyászati és Allergológiai Magánrendelés, Szolnok, Jász-Nagykun-Szolnok
  - Qualiclinic Kft, Budapest, Pest County
  - UNOMEDICALTRIALS Kft, Budapest, Pest County
- Latvia (3):
  - Riga 1st hospital, Clinic of Dermatology and STD, Riga, Rga
  - J.Kisis LtD, Riga, Rga
  - Smite Aija doctor practice in dermatology, venereology, Talsi
- Poland (16):
  - Centrum Medyczne ALL-MED Badania Kliniczne, Krakow, Maopolskie
  - Centrum Medyczne Plejady, Krakow, Maopolskie
  - MICS Centrum Medyczne Warszawa, Warsaw, Masovian Voivodeship
  - RENEW CLINIC Spolka Jawna, Bialystok
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Centrum Medyczne PROMED, Krakow
  - Barbara Rewerska Diamond Clinic, Krakow
  - ETG Siedlce, Siedlce
  - RCMed Oddzial Sochaczew, Sochaczew
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - RCMed Oddzia Warszawa, Warsaw
  - Centrum Medyczne Evimed, Warsaw
  - DermMedica Sp. z o.o., Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 87 study centers in 8 countries, including Canada, Estonia, Georgia, Germany, Hungary, Latvia, Poland, and the United States, and participated from 24 March 2021 to 28 February 2023.
Pre-assignment Details: Participants with moderate to severe plaque psoriasis were randomized at week 28 to 1 of 2 treatment groups following a run-in period. Randomization was stratified by prior biologic use for psoriasis at baseline, geographic region, and body weight group at baseline. Dosage was weight-based to ensure similar concentration by body weight received.
Groups:
- Run-in: Ustekinumab Reference Product (RP): Participants received ustekinumab RP 45 mg (baseline body weight ≤ 100 kg) or 90 mg (baseline body weight > 100 kg) on day 1 (week 0), week 4, and week 16. At week 28, eligible participants with a 50% improvement in Psoriasis Area and Severity Index (PASI 50) response or better were randomized to the continued use group (ustekinumab RP) or the switching group (ustekinumab RP and ABP 654).
- Post-randomization Switching: Ustekinumab RP and ABP 654: At week 28, eligible participants with a PASI 50 response or better were randomized to the switching group and received ABP 654 at week 28, ustekinumab RP at week 40, and ABP 654 at week 52. Ustekinumab RP and ABP 654 (45 mg [baseline body weight ≤ 100 kg] or 90 mg [baseline body weight > 100 kg]) were administered by SC injection using a pre-filled syringe.
- Post-randomization Continued-use: Ustekinumab RP: At week 28, eligible participants with a PASI 50 response or better were randomized to the continued-use group to receive ustekinumab RP 45 mg (baseline body weight ≤ 100 kg) or 90 mg (baseline body weight > 100 kg) at weeks 28, 40, and 52. Ustekinumab RP was administered by SC injection using a pre-filled syringe.
Period: Run-in Period
Arm/Group | Run-in: Ustekinumab Reference Product (RP) | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP
Started | 494 | 0 | 0
Completed | 453 | 0 | 0
Not Completed | 41 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Required alternative therapy | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Abnormal liver function | 1 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0
Not completed — Did not meet PASI 50 | 15 | 0 | 0
Not completed — Study site closure | 2 | 0 | 0
Not completed — Pregnancy | 2 | 0 | 0
Period: Post-randomization Period
Arm/Group | Run-in: Ustekinumab Reference Product (RP) | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP
Started | 0 | 228 | 225
Full Analysis Set | 0 | 228 | 225
Safety Analysis Set | 0 | 228 | 224
Completed | 0 | 209 | 209
Not Completed | 0 | 19 | 16
Not completed — Military service | 0 | 1 | 0
Not completed — Adverse Event | 0 | 4 | 2
Not completed — Lost to Follow-up | 0 | 6 | 6
Not completed — Withdrawal by Subject | 0 | 7 | 6
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Study site closure | 0 | 0 | 1
Not completed — Family planning | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the full analysis set which included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP | Total
Number analyzed (Participants) | 228 | 225 | 453
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (13.36) | 48.1 (13.48) | 47.5 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 83 | 147
  Male | 164 | 142 | 306
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 23 | 49
  Not Hispanic or Latino | 202 | 201 | 403
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 207 | 214 | 421
  Asian | 9 | 3 | 12
  Black or African American | 7 | 1 | 8
  Other | 3 | 2 | 5
  American Indian or Alaska Native | 1 | 2 | 3
  Native Hawaiian or other Pacific Islander | 1 | 2 | 3
  Not allowed to collect | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) Over the Dosing Interval (AUCtau) Between Week 52 and Week 64
Description: AUCtau from time 0 (week 52) over the dosing interval up to week 64 is presented. Pharmacokinetic (PK) parameters are based on ABP 654 in the switching group and on ustekinumab in the continued-use group.
Time Frame: Blood samples were taken pre-dose week 52; and at 2 days, 7 days, 10 days, 2 weeks, 4 weeks, 8 weeks, and 12 weeks after the week 52 dose
Population: The PK parameter analysis set consisted of all randomized participants who received all 3 doses of the assigned investigational product between week 28 and week 52 and who had an evaluable ABP 654 or ustekinumab serum concentration-time profile between week 52 and week 64. Participants with data available are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*mcg/mL
Arm/Group | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP
Number analyzed (Participants) | 199 | 204
hour*mcg/mL | 5144.40 (45.3) | 5768.45 (50.4)
Statistical Analysis 1: Comparison: Post-randomization Switching: Ustekinumab RP and ABP 654 vs Post-randomization Continued-use: Ustekinumab RP; The ratio of geometric LS means, and 90% confidence intervals (CIs) were estimated using the analysis of covariance (ANCOVA) model adjusted for the actual stratification factors if prior biologic use for psoriasis, baseline body weight group, geographic region, and PK trough concentration at week 28; Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Geometric Least Squares (LS) Means Ratio = 0.9325, 90% CI 2-sided [0.8874 to 0.9799] — Switching group vs Continued-use group

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax) Between Week 52 and Week 64
Description: Cmax between week 52 and week 64 is presented. PK parameters are based on ABP 654 in the switching group and on ustekinumab in the continued-use group.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP
Number analyzed (Participants) | 204 | 205
mcg/mL | 5.78 (41.4) | 6.31 (46.8)
Statistical Analysis 1: Comparison: Post-randomization Switching: Ustekinumab RP and ABP 654 vs Post-randomization Continued-use: Ustekinumab RP; The ratio of geometric LS means, and 90% CIs were estimated using the ANCOVA model adjusted for the actual stratification factors if prior biologic use for psoriasis, baseline body weight group, geographic region, and PK trough concentration at week 28; Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Geometric LS Means Ratio = 0.9483, 90% CI 2-sided [0.8977 to 1.0018] — Switching group vs Continued-use group

3. Secondary Outcome: Time of Maximum Serum Concentration (Tmax) Between Week 52 and Week 64
Description: Tmax between week 52 and week 64 is presented. PK parameters are based on ABP 654 in the switching group and on ustekinumab in the continued-use group.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP
Number analyzed (Participants) | 204 | 205
hours | 167.80 [41.4 to 355.2] | 168.93 [43.6 to 407.6]

4. Secondary Outcome: Serum Trough Concentration at Steady-state (Ctrough,ss) at Week 28, Week 40, and Week 52
Description: Ctrough,ss at weeks 28, 40, and 52 are presented. PK parameters are based on ABP 654 in the switching group and on ustekinumab in the continued-use group.
Time Frame: Blood samples were taken pre-dose week 28, week 40, and week 52
Population: The PK parameter analysis set consisted of all randomized participants who received all 3 doses of the assigned investigational product between week 28 and week 52 and who had an evaluable ABP 654 or ustekinumab serum concentration-time profile between week 52 and week 64. Participants with data available at each time point are presented and all participants in the overall number of participants analyzed contributed to the data in the endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP
Number analyzed (Participants) | 204 | 205
ng/mL
  Week 28: number analyzed (Participants) | 194 | 198
  Week 28 | 570.46 (105.9) | 595.86 (110.0)
  Week 40: number analyzed (Participants) | 193 | 200
  Week 40 | 537.52 (96.4) | 590.61 (103.9)
  Week 52: number analyzed (Participants) | 196 | 201
  Week 52 | 562.51 (114.0) | 599.11 (108.5)
Statistical Analysis 1: Comparison: Post-randomization Switching: Ustekinumab RP and ABP 654 vs Post-randomization Continued-use: Ustekinumab RP; The ratio of Geometric LS means, and 90% CI for Ctrough,ss at week 28 were estimated based on an ANCOVA model adjusted for the actual stratification factors of prior biologic use for psoriasis, baseline body weight group, and geographic region; Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Geometric LS Means Ratio = 0.9617, 90% CI 2-sided [0.8319 to 1.1119] — Ctrough,ss at Week 28: Switching group vs Continued-use group
Statistical Analysis 2: Comparison: Post-randomization Switching: Ustekinumab RP and ABP 654 vs Post-randomization Continued-use: Ustekinumab RP; The ratio of geometric LS means, and 90% CI for Ctrough,ss at week 40 between the 2 treatment groups were estimated using an ANCOVA model adjusting for stratification factors and PK trough concentration at week 28; Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Geometric LS Means Ratio = 0.9662, 90% CI 2-sided [0.8879 to 1.0515] — Ctrough,ss at Week 40: Switching group vs Continued-use group
Statistical Analysis 3: Comparison: Post-randomization Switching: Ustekinumab RP and ABP 654 vs Post-randomization Continued-use: Ustekinumab RP; The ratio of geometric LS means, and 90% CI for Ctrough,ss at week 52 between the 2 treatment groups were estimated using an ANCOVA model adjusting for stratification factors and PK trough concentration at week 28; Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Geomtric LS Means Ratio = 0.9806, 90% CI 2-sided [0.8916 to 1.0785] — Ctrough,ss at Week 52: Switching group vs Continued-use group

5. Secondary Outcome: PASI Percent Improvement From Baseline at Week 64
Description: The PASI is a measure of the average redness (erythema), thickness (induration), and scaliness (scaling), each graded on a 0 to 4 scale of the lesions, weighted by the area of involvement. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). PASI percent improvement is defined as 100 x (value at baseline - value at post-baseline visit) / value at baseline. A positive value indicates PASI improvement. Baseline data were derived based on observed data and at week 64 were derived based on multiple imputation (MI) data. Baseline was defined as the last non-missing assessment taken prior to the first dose of investigational product for the study.
Time Frame: Baseline (day 1) and week 64
Population: The per-protocol efficacy analysis set included all participants who were randomized and received all 3 doses of the assigned interventional product between week 28 and week 52 and who did not experience an important protocol deviation during the study that could affect the evaluation of the efficacy endpoints. The overall number of participants analyzed includes those imputed by MI as well as those with observed data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP
Number analyzed (Participants) | 216 | 215
Percentage change | 88.80 (18.066) | 88.72 (16.128)
Statistical Analysis 1: Comparison: Post-randomization Switching: Ustekinumab RP and ABP 654 vs Post-randomization Continued-use: Ustekinumab RP; Multiple imputation was applied for the point estimate and CI of the mean difference between the switching and continued-use groups. Missing PASI scores at the week 64 visit were imputed by MI; Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Mean difference = 0.07, 90% CI 2-sided [-2.62 to 2.77] — Mean difference in PASI percent improvement from baseline at Week 64: Switching group - Continued-use group

6. Secondary Outcome: PASI 75 Response at Week 64
Description: The PASI is a measure of the average redness (erythema), thickness (induration), and scaliness (scaling), each graded on a 0 to 4 scale of the lesions, weighted by the area of involvement. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). PASI response was defined as a participant meeting or surpassing a pre-specified threshold for percent improvement in PASI score compared to the baseline PASI score. An improvement of at least 75% qualified a participant as being a PASI 75 responder. Missing PASI 75 responses at week 64 were imputed by non-responder imputation (NRI). Baseline was defined as the last non-missing assessment taken prior to the first dose of investigational product for the study.
Time Frame: Baseline (day 1) and week 64
Population: The per-protocol efficacy analysis set included all participants who were randomized and received all 3 doses of the assigned interventional product between week 28 and week 52 and who did not experience an important protocol deviation during the study that could affect the evaluation of the efficacy endpoints. The overall number of participants analyzed includes those imputed by NRI as well as those with observed data.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP
Number analyzed (Participants) | 216 | 215
Percentage of responders | 83.3 [78.4 to 88.3] | 82.8 [77.8 to 87.8]
Statistical Analysis 1: Comparison: Post-randomization Switching: Ustekinumab RP and ABP 654 vs Post-randomization Continued-use: Ustekinumab RP; Response difference was estimated by the Mantel-Haenszel estimate, and the 90% CIs were estimated by the stratified Newcombe confidence limits, adjusting for the prior biologic use of psoriasis, baseline body weight group, geographic region. Missing post-baseline binary response data were imputed by NRI; Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Response difference = 0.2, 90% CI 2-sided [-5.7 to 6.2] — Response difference in PASI 75 Response at Week 64: Switching group - Continued-use group

7. Secondary Outcome: PASI 100 Response at Week 64
Description: The PASI is a measure of the average redness (erythema), thickness (induration), and scaliness (scaling), each graded on a 0 to 4 scale of the lesions, weighted by the area of involvement. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). PASI response was defined as a participant meeting or surpassing a pre-specified threshold for percent improvement in PASI score compared to the baseline PASI score. An improvement of 100% qualified a participant as being a PASI 100 responder. Missing PASI 100 responses at week 64 were imputed by NRI. Baseline was defined as the last non-missing assessment taken prior to the first dose of investigational product for the study.
Time Frame: Baseline (day 1) and week 64
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP
Number analyzed (Participants) | 216 | 215
Percentage of responders | 36.1 [29.7 to 42.5] | 35.8 [29.4 to 42.2]
Statistical Analysis 1: Comparison: Post-randomization Switching: Ustekinumab RP and ABP 654 vs Post-randomization Continued-use: Ustekinumab RP; [analysis description as in outcome 6, analysis 1]; Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Response difference = 0.2, 90% CI 2-sided [-7.4 to 7.8] — Response difference in PASI 100 Response at Week 64: Switching group - Continued-use group

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs): Post-randomization Period
Description: TEAEs during the post-randomization period were defined as AEs that started on or after the first dose of investigational product post-randomization and prior to the end of study. The number of participants who experienced any TEAE, and who experienced a serious TEAE are presented. A serious TEAE was defined as any untoward medical occurrence that meets at least 1 of the following serious criteria: resulted in death (fatal), was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly/birth defect, or other medically important serious event.
Time Frame: Week 28 to week 64
Population: The safety analysis set included all randomized participants who received at least 1 dose of investigational product post randomization.
Measure: Count of Participants; unit: Participants
Groups:
- Post-randomization Switching: Ustekinumab RP and ABP 654: Participants were randomized to the switching group at week 28 and completed all planned doses of ABP 654 and ustekinumab RP up to week 52, including ABP 654 at week 28, ustekinumab RP at week 40, and ABP 654 at week 52.
- Post-randomization Continued-use: Ustekinumab RP: Participants were randomized to the continued-use group at week 28 and completed all planned doses of ustekinumab RP up to week 52, including 3 doses at weeks 28, 40, and 52.
- Post-randomization Switching: ABP 654/Ustekinumab RP/Missing: Participants were randomized to the switching group at week 28 and received ABP 654 at week 28 and ustekinumab RP at week 40 but did not receive the planned dose of ABP 654 at week 52.
- Post-randomization Continued-use: Ustekinumab RP/Ustekinumab RP/Missing: Participants were randomized to the continued-use group at week 28 and received ustekinumab RP at week 28 and week 40 but did not receive the planned dose of ustekinumab RP at week 52.
- Post-randomization Switching: ABP 654/Missing/Missing: Participants were randomized to the switching group at week 28 and received ABP 654 at week 28 and did not receive the planned doses of ustekinumab RP at week 40 and ABP 654 at week 52.
- Post-randomization Continued-use: Ustekinumab RP/Missing/Missing: Participants were randomized to the continued-use group at week 28 and received ustekinumab RP at week 28 but did not receive the planned doses of ustekinumab RP at week 40 and week 52.
Arm/Group | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP | Post-randomization Switching: ABP 654/Ustekinumab RP/Missing | Post-randomization Continued-use: Ustekinumab RP/Ustekinumab RP/Missing | Post-randomization Switching: ABP 654/Missing/Missing | Post-randomization Continued-use: Ustekinumab RP/Missing/Missing
Number analyzed (Participants) | 217 | 216 | 8 | 5 | 3 | 3
Participants
  Any TEAE | 97 | 108 | 4 | 1 | 3 | 0
  Any serious TEAE | 3 | 2 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Events of Interest (EOI): Post-randomization Period
Description: The treatment-emergent EOIs prespecified for this study included serious systemic hypersensitivity reactions, facial palsy, pustular psoriasis, erythrodermic psoriasis, serious infections (including mycobacterial and salmonella infections), malignancy, cardiovascular events, reversible posterior leukoencephalopathy syndrome (RPLS), serious depression including suicidality, and venous thromboembolism.
Time Frame: Week 28 to week 64
Population: Participants in the safety analysis set who completed all planned doses of investigational product in the post-randomization period up to week 52. The safety analysis set included all randomized participants who received at least 1 dose of investigational product post randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP
Number analyzed (Participants) | 217 | 216
Participants
  Any EOI | 6 | 7
  Cardiovascular events | 2 | 3
  RPLS | 2 | 0
  Serious infections | 1 | 2
  Malignancy | 1 | 1
  Serious depression | 0 | 1
  Serious systemic hypersensitivity reactions | 0 | 0
  Facial palsy | 0 | 0
  Pustular psoriasis | 0 | 0
  Erythrodermic psoriasis | 0 | 0
  Venous thromboembolism | 0 | 0
Statistical Analysis 1: Comparison: Post-randomization Switching: Ustekinumab RP and ABP 654 vs Post-randomization Continued-use: Ustekinumab RP; Risk difference for any EOI: risk difference and CIs were estimated by Wald asymptotic confidence limits, or exact confidence limits if n < 25 for either treatment; Test type: Equivalence — The prespecified similarity margin was 0.8 to 1.25; Risk Difference (RD) = -0.48, 90% CI 2-sided [-4.17 to 3.10] — Switching group - continued-use group

10. Secondary Outcome: Number of Participants With Antidrug Antibodies (ADAs): Post-randomization Period
Description: The number of participants developing binding or neutralizing ADAs during the post-randomization period is defined as the number of participants in the safety analysis set who had a positive result post-randomization and had never tested positive (i.e., negative or no results) prior to the first dose of post-randomization investigational product and who have at least one ADA result post randomization. A transient antibody results was defined as a positive result during the post-randomization period with a negative result at the participant's last visit tested within the respective study period. Baseline was defined as the last non-missing assessment taken prior to the first dose of investigational product for the study.
Time Frame: Baseline (pre-dose day 1), week 4, week 16, week 28, week 40, week 52 and week 64
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP | Post-randomization Switching: ABP 654/Ustekinumab RP/Missing | Post-randomization Continued-use: Ustekinumab RP/Ustekinumab RP/Missing | Post-randomization Switching: ABP 654/Missing/Missing | Post-randomization Continued-use: Ustekinumab RP/Missing/Missing
Number analyzed (Participants) | 217 | 216 | 8 | 5 | 3 | 3
Participants
  Participants with post-baseline result post-randomization | 217 | 216 | 8 | 5 | 3 | 1
  Binding antibody negative/no result prior to first dose post-randomization | 136 | 134 | 5 | 4 | 3 | 1
  Binding antibody positive with negative/no result prior to first dose post-randomization | 7 | 11 | 0 | 1 | 1 | 0
  Transient binding antibody positive with negative/no result prior to first dose post-randomization | 4 | 5 | 0 | 0 | 0 | 0
  Neutralizing antibody negative/no result prior to first dose post-randomization | 190 | 188 | 6 | 5 | 3 | 1
  Neutralizing antibody positive with negative/no result prior to first dose post-randomization | 8 | 6 | 0 | 1 | 0 | 0
  Transient neutralizing antibody positive with negative/no result prior first dose post-randomization | 6 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from enrollment to the end of study visit, up to approximately 68 weeks. Adverse events were collected from Day 1 to end of study, up to 64 weeks.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Run-in: Ustekinumab RP: Participants received ustekinumab RP 45 mg (baseline body weight ≤ 100 kg) or 90 mg (baseline body weight > 100 kg) on day 1 (week 0), week 4, and week 16.
Arm/Group | Run-in: Ustekinumab RP | Post-randomization Switching: Ustekinumab RP and ABP 654 | Post-randomization Continued-use: Ustekinumab RP | Post-randomization Switching: ABP 654/Ustekinumab RP/Missing | Post-randomization Continued-use: Ustekinumab RP/Ustekinumab RP/Missing | Post-randomization Switching: ABP 654/Missing/Missing | Post-randomization Continued-use: Ustekinumab RP/Missing/Missing
All-Cause Mortality (participants affected / at risk) | 2/494 | 0/217 | 0/216 | 0/8 | 0/5 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 14/494 | 3/217 | 2/216 | 0/8 | 0/5 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 116/494 | 55/217 | 58/216 | 4/8 | 1/5 | 3/3 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in: Ustekinumab RP (N=494) | Post-randomization Switching: Ustekinumab RP and ABP 654 (N=217) | Post-randomization Continued-use: Ustekinumab RP (N=216) | Post-randomization Switching: ABP 654/Ustekinumab RP/Missing (N=8) | Post-randomization Continued-use: Ustekinumab RP/Ustekinumab RP/Missing (N=5) | Post-randomization Switching: ABP 654/Missing/Missing (N=3) | Post-randomization Continued-use: Ustekinumab RP/Missing/Missing (N=3)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatillomania (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in: Ustekinumab RP (N=494) | Post-randomization Switching: Ustekinumab RP and ABP 654 (N=217) | Post-randomization Continued-use: Ustekinumab RP (N=216) | Post-randomization Switching: ABP 654/Ustekinumab RP/Missing (N=8) | Post-randomization Continued-use: Ustekinumab RP/Ustekinumab RP/Missing (N=5) | Post-randomization Switching: ABP 654/Missing/Missing (N=3) | Post-randomization Continued-use: Ustekinumab RP/Missing/Missing (N=3)
COVID-19 (Infections and infestations) | 65 | 27 | 25 | 2 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 27 | 12 | 16 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 6 | 1 | 3 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 18 | 14 | 14 | 0 | 0 | 0 | 0
Abdominal wall wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 1 | 1 | 0
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 9 | 5 | 1 | 0 | 1 | 0 | 0
Scleroedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT04761627/Prot_002.pdf
  • Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT04761627/SAP_003.pdf